CLINICAL TRIAL: NCT03970772
Title: Mini-Dose Glucagon to Treat Fasting-induced Hypoglycemia During Ramadan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qassim University (Other)
Responsible Party: Principal Investigator, Metab Algeffari, Associate Professor, Diabetologist Consultant, Qassim University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: med-2019-2-2-I-5389
Record Dates: First submitted 2019-05-29; First posted 2019-06-03 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Fasting Hypoglycemia; Diabetes Mellitus, Type 1
Keywords: Type 1 diabetes mellitus; Fasting; Ramadan; Glucagon; Mini-dose; Hypoglycemia
MeSH Terms: conditions — Hypoglycemia; Diabetes Mellitus, Type 1; Fasting | interventions — Glucagon; Glucose

STUDY DESIGN:
Intervention Model Description: This is a Randomize Crossover study with a pre-crossover phase and a crossover trial phase, which will include a minimum of 20 participants and consist of two (2-weeks) periods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glucagon injection (Experimental): Dilute Glucagon (1 mg/ml)
  Interventions: Drug: Glucagon Injection
- Glucose tablets (Active Comparator): Dextrose glucose tablets
  Interventions: Other: Glucose Tablets

INTERVENTIONS:
Drug: Glucagon Injection — Participants will be instructed to check their blood glucose (BG) with study meter once they developed hypoglycemia symptoms, their CGM reads below 70 mg/dl, or when the CGM glucose was trending down and the participant intended to treat to prevent hypoglycemia. Participants will be instructed to check BG with meter 3 times and treat the hypoglycemia event using mini-dose glucagon when their BG in range 40-69 mg/dl according a prescribed protocol.
  Arms: Glucagon injection
Other: Glucose Tablets — Participants will be instructed to check their blood glucose (BG) with study meter once they developed hypoglycemia symptoms, their CGM reads below 70 mg/dl, or when the CGM glucose was trending down and the participant intended to treat to prevent hypoglycemia. Participants will be instructed to check BG with meter 3 times and treat the hypoglycemia event using glucose tablets when their BG in range 40-69 mg/dl according a prescribed protocol.
  Arms: Glucose tablets

SUMMARY:
This study aimed to develop a new approach for the treatment of fasting induced hypoglycemia during ramadan using mini-dose glucagon.

DETAILED DESCRIPTION:
This study aimed to understand whether subcutaneously-given mini-dose glucagon (MDG) as an alternative to carbohydrate consumption could avert hypoglycemia or treat it effectively in type 1 diabetes patients who choose to fast during Ramadan in observance of their faith. This treatment method could also avert any negative psychological emotions Muslim people with diabetes may experience by ingesting carbohydrates to control hypoglycemia, thereby breaking their fast. Furthermore, it could improve ability to self-manage fasting, which is an important action for their spiritual and overall wellbeing.

There will be two phases included in this study:

1. Pre-crossover Phase:

   Before starting the crossover trial, a pre-crossover phase will conduct to evaluate hypoglycemia eligibility, frequency and compliance.
2. Crossover Trial Phase:

The Crossover Trial Phase will include 20 participants and consist of two (2-weeks) periods. Participants who don't develop any hypoglycemic event or failed to complete both periods will be excluded.

Participants will be randomized into two groups:

1. Group A in periods one will use MDG and glucose tablets in period two according to the protocol.
2. Group B in periods one will use glucose tablets and MDG in period two according to the protocol.

The primary outcome will be the number of treated fasting induced hypoglycemic events.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of T1DM using daily insulin
2. 18.0 to < 65.0 years of age with body mass index 20.0 to <35.0 kg/m2.
3. Having diabetes for ≥2.0 years
4. HbA1c <8.5%
5. Has a smart phone with access to the internet and welling to upload data during the study period.
6. Welling to wear a devise such as continuous glucose monitor ≥6 days/week.
7. Females, not currently known to be pregnant
8. In good general health as evaluated by investigator based on available clinical data
9. Willing to comply to the protocol requirements for the duration of the study

Exclusion Criteria:

1. Any history of more than one severe hypoglycemic episode (need assistance by third party) in the past 12 months
2. Any history of more than one episode of diabetic ketoacidosis in the past 12 months
3. Female pregnant or planning to get pregnant.
4. Use of any of the following medications: oral hypoglycemic agents, systemic corticosteroids or beta-blocker, theophylline, beta-adrenergic agonists, 1st generation anticholinergic drugs.
5. History of hypersensitivity to glucagon or severe hypersensitivity reactions (such as angioedema) to any other medications
6. History of uncontrolled hypertension (systolic BP >160 mmHg or diastolic BP >100 mmHg)
7. History of seizure disorder.
8. Presence of any of conditions based on judgment of the investigator that could affect or interfere with the response, absorption, metabolism or execration of glucagon.
9. Currently following any kind of weight-loss diet
10. Currently participation in another clinical trials

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-08-15 (Actual)

PRIMARY OUTCOMES:
Changes in glucose values from baseline to 30 minute | 30 minutes
  The change in blood glucose from baseline to 30 minute following treatment of hypoglycemic events

SECONDARY OUTCOMES:
Events approached 100 mg/dL or increased by 30 mg/dL | 60 Minutes
  During the first hour following each hypoglycemic event (BG 50-69 mg/dL), the investigators will record the events approached 100 mg/dL or increased by 30 mg/dL
Treatment success from first dose | 60 Minutes
  During the first hour following each hypoglycemic event (BG 50-69 mg/dL), the investigators will record the events with blood glucose concentration ≥50 mg/dl 15 minute AND ≥70 mg/dl 30 minute after the initial treatment of a hypoglycemic event
Mean Glucose Value, during hypoglycemia event by CGM | 60 Minutes
  During the first hour following each hypoglycemic event (BG 50-69 mg/dL), the investigators will calculate the mean glucose value from CGM data
Time in Range, during hypoglycemia event by CGM | 60 Minutes
  During the first hour following each hypoglycemic event (BG 50-69 mg/dL), the investigators will calculate the percentage of time in range 70-180 mg/dL from CGM data.
Time spend below 70 mg/dL, during hypoglycemia event by CGM | 60 Minutes
  During the first hour following each hypoglycemic event (BG 50-69 mg/dL), the investigators will calculate the percentage of time <70 mg/dL from CGM data.
Minimum Glucose, during hypoglycemia event by CGM | 60 Minutes
  During the first two hour following each hypoglycemic event (BG 50-69 mg/dL), the investigators will record the minimum glucose value from CGM data.
Maximum Glucose, during hypoglycemia event by CGM | 60 Minutes
  During the first two hour following each hypoglycemic event (BG 50-69 mg/dL), the investigators will record the maximum glucose value from CGM data.
Mean Glucose Value, during hypoglycemia event by CGM | 120 Minutes
  During the first two hour following each hypoglycemic event (BG 50-69 mg/dL), the investigators will calculate the mean glucose value from CGM data
Time in Range, during hypoglycemia event by CGM | 120 Minutes
  During the first two hour following each hypoglycemic event (BG 50-69 mg/dL), the investigators will calculate the percentage of time in range 70-180 mg/dL from CGM data
Time spend below 70 mg/dL, during hypoglycemia event by CGM | 120 Minutes
  During the first two hour following each hypoglycemic event (BG 50-69 mg/dL), the investigators will calculate the percentage of time <70 mg/dL from CGM data
Minimum Glucose, during hypoglycemia event by CGM | 120 Minutes
  During the first two hour following each hypoglycemic event (BG 50-69 mg/dL), the investigators will record the minimum glucose value from CGM data.
Maximum Glucose, during hypoglycemia event by CGM | 120 Minutes
  During the first two hour following each hypoglycemic event (BG 50-69 mg/dL), the investigators will record the maximum glucose value from CGM data.
The proportion of completion of fasts | 2 Weeks
  The proportion of completion of fasts following treatment of hypoglycemic events
Mean Glucose Value, by CGM | 2 Weeks
  During the entire two weeks of intervention/comparator period, the investigators will calculate the mean glucose value from CGM data
Time in Range, by CGM | 2 Weeks
  During the entire two weeks of intervention/comparator period, the investigators will calculate the percentage of time in range 70-180 mg/dL from CGM data
Time spend below 70 mg/dL, by CGM | 2 Weeks
  During the entire two weeks of intervention/comparator period, the investigators will calculate the percentage of time <70 mg/dL from CGM data
Time spend above 180 mg/dL, by CGM | 2 Weeks
  During the entire two weeks of intervention/comparator period, the investigators will calculate the percentage of time >180 mg/dL from CGM data
Time spend above 250 mg/dL, by CGM | 2 Weeks
  During the entire two weeks of intervention/comparator period, the investigators will calculate the percentage of time >250 mg/dL from CGM data
Coefficient of Variation, by CGM | 2 Weeks
  During the entire two weeks of intervention/comparator period, the investigators will calculate the Coefficient of Variation from CGM data

CONTACTS AND LOCATIONS:
Locations (1):
- Qassim University, Buraidah, Saudi Arabia

REFERENCES:
- [Derived] Algeffari M, Hussain S, Almogbel T, Alsharidah M, Alghadouni H, Mahmood F. Home Use of Mini-Dose Glucagon As a Novel Treatment for Hypoglycemia Following Repeated, Prolonged Fasts in Type 1 Diabetes During Ramadan. Diabetes Care. 2022 Apr 1;45(4):990-993. doi: 10.2337/dc21-1655. PMID 35176134